CLINICAL TRIAL: NCT06354985
Title: Modafinil and Exercise for Post Stroke Fatigue (MODEX)
Brief Title: Modafinil and Exercise for Post Stroke Fatigue
Acronym: MODEX
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-5996; MODEX2023 (Other: Clinical Trial Protocol Number); FRN:183960 (Other Grant/Funding Number: CIHR); CTO Project ID: 4701 (Other: Clinical Trials Ontario)
Record Dates: First submitted 2024-03-22; First posted 2024-04-09 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Fatigue; Modafinil; Exercise
MeSH Terms: conditions — Stroke; Fatigue; Motor Activity | interventions — Modafinil; Sugars; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All members of the research team and the participants will be blinded to medication group allocation. The study statistician who is unblinded and the Data Safety Monitoring Board will have access to the medication assignment if needed (e.g. adverse drug reaction).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Drug + Exercise (Placebo Comparator): Placebo Drug + Exercise for 8 weeks.
  Interventions: Drug: Placebo; Behavioral: Exercise
- Modafinil 200 mg/day + Exercise (Active Comparator): Modafinil 200 mg/day + Exercise for 8 weeks.
  Interventions: Drug: Modafinil 200mg; Behavioral: Exercise

INTERVENTIONS:
Drug: Modafinil 200mg — Modafinil 200mg daily for 8 weeks.
  Other Names: Modafinil
  Arms: Modafinil 200 mg/day + Exercise
Drug: Placebo — Placebo daily for 8 weeks.
  Other Names: Sugar Pill
  Arms: Placebo Drug + Exercise
Behavioral: Exercise — Exercise three times per week for 8 weeks.

SUMMARY:
A stroke happens when blood flow to the brain is stopped and the brain gets damaged. At least half of people with a stroke have fatigue months and even years later. A lot of people report fatigue as one of the worst symptoms post stroke that can affect daily activities and the length and quality of life. Though all the reasons for fatigue after stroke and how to best treat it are not fully understood, the investigators think that fatigue results from the stroke changing the brain, reducing physical fitness, and decreasing muscle strength. A stroke can also affect sleep and mood, which can impact how people feel too. It is also not known why women experience more fatigue than men after a stroke.

Some studies have tested a drug called Modafinil for post stroke fatigue, while other studies have tested exercise for it. Yet, there is unclear evidence for either treatment, so this study has the following aim:

1. Test if Exercise plus Modafinil is better than Exercise plus a Sugar Pill

This study will take place at up to 6 Canadian research sites to give a good representation of people after a stroke. Each person will be tested on fatigue, mood, fitness, thinking skills, sleep, and usual activity levels.

Participants will be assigned at random (like flipping a coin) to 1 of 2 groups:

1. Sugar Pill plus Exercise
2. Modafinil plus Exercise

The treatment will last 8 weeks. The Modafinil or Sugar Pill will be taken once a day. The exercise will be delivered virtually by a trained therapist over computer to people at home 3 times a week. Change in fatigue, quality of life, and other outcomes will be measured over 6 months.

The investigators will assess the results to identify the best treatment for post stroke fatigue and hope to be able to find a treatment that will help reduce fatigue and improve quality of life after a stroke.

DETAILED DESCRIPTION:
Study Rationale Post stroke fatigue (PSF) afflicts as many as 70% of the 400,000 Canadians with stroke. People with stroke endorse PSF as the most serious unmet research priority. Pathological fatigue is not relieved by rest and is characterized by persistent or extreme tiredness, exhaustion, and/or difficulty in initiating or sustaining voluntary activities. PSF is an excellent exemplar to study as the cause of disabling PSF is unclear. Systematic reviews confirm that PSF is multifactorial having both peripheral (e.g. cardiovascular and neuromuscular) and central (e.g. alterations in brain function resulting in both physical and psychological symptoms) components. There are no evidence-based treatments for PSF, however, exercise and the dopaminergic medication Modafinil that targets the dopaminergic movement circuits in the brain, have shown promise in alleviating symptoms in small studies.

Study Design This multicentre clinical trial will involve a double blind randomized controlled trial design to quantify the effect of a structured exercise program combined with Modafinil 200 mg daily or placebo medication over 8 weeks on severity of fatigue symptoms. It aims to recruit 212 participants into one of two arms. It will also explore the interactions of Modafinil in combination with exercise. The effects of mood, sleep, stroke impairments, sex, gender and activity levels on post stroke fatigue will also be explored.

Study Population Study participants must meet the inclusion/exclusion criteria at the time of entry into the study. In general, participants will be >3 months post stroke onset (i.e. intracerebral hemorrhage or ischemic stroke diagnosed by a physician) at the time of consent into the study.

Primary Hypothesis The primary hypothesis based on outcomes at 8 weeks is that structured telerehabilitation fitness and strengthening exercise plus Modafinil will improve fatigue symptom severity more than placebo medication and the same exercise.

ELIGIBILITY:
Inclusion Criteria

1. >18 years of age (on date of consent)
2. >3 months post stroke onset (i.e. intracerebral hemorrhage or ischemic stroke diagnosed by a physician) (on date of consent)
3. evidence of stroke on computed tomography (CT) or magnetic resonance imaging (MRI)
4. disabling post stroke fatigue as measured by Multidimensional Fatigue Inventory score >60
5. Modified Rankin disability score <4
6. Able to participate in moderate exercise for an hour (with one person assistance or less)

Exclusion Criteria

1. contraindications to Modafinil
2. on stimulant medications already
3. subarachnoid hemorrhage
4. impaired comprehension or language impairment that prevents following visual or pictograph adapted instructions or providing informed consent
5. severe motor impairment or inability to participate in the exercise
6. unable to participate in exercise due to musculoskeletal complaints, unstable heart failure, or renal disease
7. untreated hypothyroidism or anemia
8. cancer likely to result in death in <6 months
9. severe depression requiring therapy as indicated by suicidal ideation and/or Depression Anxiety Stress Scales (DASS) depression sub-score >20
10. currently enrolled in a structured exercise program
11. untreated severe sleep apnea with an Apnea/Hypopnea index >30 as measured by validated wearable sleep apnea detector
12. pregnant, breastfeeding, or positive test for pregnancy at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Severity of Fatigue Symptoms | Week 8
  Multidimensional Fatigue Inventory

SECONDARY OUTCOMES:
Severity of Fatigue Symptoms | Week 4 and 26
  Multidimensional Fatigue Inventory
Impact on Quality of Life | Week 8 and 26
  Medical Outcomes Short Form Scale
Walking Recovery | Week 8 and 26
  Timed Up and Go
Leg Strength and Coordination | Week 8 and 26
  30-Second Sit to Stand Test
3-Day Physical Activity Assessment | Week 8
  Activity Accelerometer
Mood and Anxiety | Week 4, 8, and 26
  Depression Anxiety Stress Scales
Attention | Week 8 and 26
  Montreal Cognitive Assessment
Cognition | Week 8 and 26
  Trails Tests
Health Resource Utilization | Week 4, 8, and 26
  Health Resource Utilization Questionnaire
Quality Adjusted Life Years | Week 4, 8, and 26
  Cost Per Quality Adjusted Life Years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bayley, MD, FRCPC, Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: No